CLINICAL TRIAL: NCT06056622
Title: Overcoming Motion Sickness in Immersive Virtual Reality
Brief Title: Motion Sickness Rehabilitation for Virtual Reality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Ramazan KURUL, Assist. Prof, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AIBU-FTR-RK-07
Record Dates: First submitted 2023-09-21; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Motion Sickness
Keywords: Rehabilitation; Balance; Reflex
MeSH Terms: conditions — Motion Sickness

STUDY DESIGN:
Intervention Model Description: Two groups with a sham control. Assessments will be performed before intervention, and four months after the last session.
Who Masked: Participant, Outcomes Assessor
Masking Description: The intervention group will receive combined exercise program and the control group will receive a sham exercise using reaction time games. Outcome assessment will be performed by an investigator who was unaware of group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined Exercise Group (Other): Multisensory stimulation with active range of motion movement, progressive Cawthorne-Cooksey exercises, and balance exercises with external perturbation on soft and hard surfaces while eyes are open or closed.
  Interventions: Other: Combined Exercises
- Control Group (Other): A placebo exercise program consist of 10 minute reaction time game which requires mouse clicking on screen color changes will be used in control group.
  Interventions: Other: Placebo Exercise

INTERVENTIONS:
Other: Combined Exercises — The treatment involving multisensory stimulation through active movement was structured into two distinct segments. The initial segment encompassed exercises executed on a wobble board, comprising tasks such as squats, passing a ball between hands and to another individual, maintaining a single-leg stance, and gently destabilizing each other's balance. The subsequent segment involved exercises performed on a soft mat, including activities such as jumping from a small box and landing with both knees flexed, passing the ball to a team member during a two-leg jump, executing a two-leg jump while rotating the trunk by 90 degrees, and leaping from a small box onto a soft mat while balancing on one leg. Each of these exercises was repeated ten times within each session.
  Balance-related exercises were conducted with participants assuming a shoulder-width stance on both firm and soft surfaces.
  Arms: Combined Exercise Group
Other: Placebo Exercise — Participants allocated to the control group will receive placebo treatment sessions, which entailed a 10-minute exposure to a visual evoked potential (VEP) measurement screen while holding a mouse. During this time, participants were given instructions to click the mouse whenever the screen exhibited a change in color. These activities were carried out while seated in a chair equipped with arm support
  Arms: Control Group

SUMMARY:
The objective of this study was to investigate the effect of a rehabilitation program on motion sickness. A combined rehabilitation program will be given participants who showed motion sickness symptoms.

DETAILED DESCRIPTION:
In the realm of virtual environments and simulators, a significant hurdle that hampers user engagement resides in the manifestation of adverse effects. These deleterious consequences become apparent during prolonged exposure to virtual settings, with approximately 30% of users grappling with symptoms like nausea and up to 40% reporting eyestrain. Furthermore, users frequently describe a constellation of other discomforting sensations, including headaches, dizziness or vertigo, compromised postural stability, drowsiness, increased salivation, and perspiration. These adverse effects have been documented in scientific literature under various monikers, with 'cybersickness' and 'motion sickness' (MS) being the most prevalent designations.

Motion sickness, a vexing symptom characterized by discomfort experienced during movements unrelated to one's bodily motions, such as those encountered during travel by air, sea, or land, lies at the crux of this issue. The pathophysiological elucidation of the mechanisms underlying MS centers around the notion of sensory conflict or sensory mismatch. This conflict arises from disparities between the sensory information derived from kinaesthetic inputs, the vestibular and visual systems, and the sensory patterns engendered by the virtual environment

ELIGIBILITY:
Inclusion Criteria:

* having stereoacuity score of 3552 arc/s on the Titmus Fly Test

Exclusion Criteria:

* having partial or total vision loss
* being diagnosed with vertigo
* having previous experience of head mounted virtual reality devices

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2022-12-04 (Actual); Primary Completion 2023-04-23 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Virtual Reality Symptoms Questionnaire | four weeks
  o gauge motion sickness symptoms, a 9-question Likert scale was employed. Participants were directed to rate the extent to which each of the specified symptoms affected them, using a scale ranging from 0 (no impact) to 3 (severe impact). The total score for this assessment totaled 100, with scores derived from two distinct subsections: oculomotor symptoms and overall discomfort.

SECONDARY OUTCOMES:
Visual Analog Scale | four weeks
  Participants were instructed to express the level of their enjoyment using a 100-millimeter horizontal line. The intensity of their experience was determined by measuring the segment on the line that the individual marked, with a scale ranging from 0 (completely unenjoyable) to 10 (the most enjoyable experience).
Biodex System Analysis | four weeks
  The Biodex System was utilized to record angular displacement of the platform in both the antero-posterior (AP) and medio-lateral (ML) axes, providing metrics for postural stability and balance. The medio-lateral stability index (MLSI) was derived from angular displacement in the frontal plane on a circular platform, while the antero-posterior stability index (APSI) was obtained from angular displacement in the sagittal plane on the same platform. The overall stability index (OSI) was calculated as a composite measure combining APSI and MLSI. During the measurements, participants were instructed to stand on the platform, either on one foot or both feet, following the prescribed protocol, and to maintain a static posture.
Flaming Balance Test | four weeks
  This test was employed to evaluate participants' static balance, with trials conducted under both eyes-closed and eyes-open conditions. Each participant was guided to place the ankle of their non-tested leg behind the knee of the tested leg while standing on one leg for a duration of 1 minute. The number of observable body sways was documented throughout the test duration.

CONTACTS AND LOCATIONS:
Overall Officials: Ramazan KURUL, PhD, Principal Investigator — Abant Izzet Baysal University
Locations (1):
- Abant Izzet Baysal University, Bolu, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
After study publication reasonable requests for systematic reviews can be accepted for detailed data sharing rest of the data will be available on online link.
Supporting Information: Study Protocol, SAP
Time Frame: Data wil lbe available after study publication and it will be available indefinitely.
Access Criteria: Data wil lbe uploaded to university's cloud servers and an online link will be shared